CLINICAL TRIAL: NCT06354491
Title: An Imaging-based Quantitative Biomarker Assay for Non-alcoholic Fatty Liver Disease (NAFLD) in Children: a Feasibility Study
Brief Title: An Imaging-based Quantitative Biomarker Assay for NAFLD in Children
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-1494; A534800 (Other: UW Madison); Protocol Version 12/19/24 (Other: UW Madison)
Record Dates: First submitted 2024-04-03; First posted 2024-04-09 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: NAFLD; NASH
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Magnetic Resonance Imaging; Ultrasonography

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Average or low BMI (Experimental): Children with BMI under the 85th percentile for age and sex
  Interventions: Device: Magnetic Resonance Imaging (MRI); Device: Ultrasound (US)
- High BMI (Experimental): Children with BMI in the 95th percentile or higher for age and sex
  Interventions: Device: Magnetic Resonance Imaging (MRI); Device: Ultrasound (US)

INTERVENTIONS:
Device: Magnetic Resonance Imaging (MRI) — MRI procedures will include a 20-25 minute exam with periodic breath holds. The imaging series will be conducted twice to assess repeatability.
Device: Ultrasound (US) — In each ultrasound exam, each participant will be scanned by twice by the same sonographer to evaluate intra-operator variability (repeatability). Each exam will take approximately 60 minutes to complete.

SUMMARY:
This study will validate recently developed Magnetic Resonance Imaging (MRI) and Ultrasound (US) based methods for liver fat quantification in children with obesity and healthy range of body mass index (BMI).

DETAILED DESCRIPTION:
The severity of the obesity epidemic in the U.S., particularly in Wisconsin, is alarming, with overall overweight or obesity rates of 35% in children. [Fryar 2020,] Obesity is a major risk factor for several comorbidities, one of the most common being non-alcoholic fatty liver disease (NAFLD, also denoted steatotic liver disease). The inflammatory state known as non-alcoholic steatohepatitis (NASH) may lead to fibrosis and, if left untreated, can lead to cirrhosis, liver failure, and cancer. For these reasons, there is enormous interest in effective interventions for weight loss and reversing NAFLD. A central challenge in the development of new interventions is the need for accurate and precise biomarkers to evaluate hepatic steatosis in children.

This pilot study focuses on demonstrating the feasibility of MRI and US based liver fat quantification in children and addresses technical challenges that may limit the performance of the proposed techniques in the population of interest through the following aims:

* Aim 1: Determine the bias and precision (repeatability) of emerging free-breathing MRI-based liver fat quantification in children with obesity and controls using current breath-held methods as a reference.
* Aim 2: Determine the precision (repeatability and reproducibility) of US-based biomarkers of liver steatosis with a focus on the impact of body wall thickness on the precision of the biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 10 - 14years old
2. BMI: Case subjects: BMI>95th percentile for age and sex Healthy BMI volunteers: 5th ≤ BMI < 85th percentile for age and sex

Exclusion Criteria:

1. Children with contraindications to MRI.
2. Children who did not fast (verbally confirmed by children or guardian)
3. Pregnant

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility Measured by the Number of Participants Who Successfully Complete the Interventions | through study enrollment (up to approximately 14 months)
  Demonstrate the feasibility of MRI- and US-based liver fat quantification in children and address technical challenges that may limit the performance of the proposed techniques in the population of interest.

SECONDARY OUTCOMES:
MRI: Bias reported as difference in mean error in Percent Liver Fat measured from free-breathing MRI method and reference breath-held MRI method | Research visit 1 (up to 14 months)
  To validate and confirm the reliability of a recently developed free-breathing CSE-based PDFF mapping method in children with high and average/low BMI for age and sex, bias is reported. Bias is defined as the mean error in liver PDFF measurements between the new free-breathing MRI method and the reference breath-held MRI method, reported in percentage.
MRI: Precision measured by Test-Retest of Percent Liver Fat | Research visit 1 (up to 14 months)
  To validate and confirm the reliability of a recently developed free-breathing CSE-based PDFF mapping method in children with high and average/low BMI for age and sex, precision will be assessed.
  Precision (test-retest repeatability) for each acquisition method and within each liver segment will be calculated through the coefficient of repeatability.
Quantitative US: Repeatability of US Measurements (same sonographer) - Attenuation Coefficient (dB/cm-MHz) | Research visit 1 (up to 14 months)
  Biomarkers of liver steatosis are measured and analyzed for their repeatability by the same sonographer in the high and healthy BMI cohorts.
Quantitative US: Repeatability of US Measurements (same sonographer) - Backscatter Coefficient (1/cm*sr) | Research visit 1 (up to 14 months)
  Biomarkers of liver steatosis are measured and analyzed for their repeatability by the same sonographer in the high and healthy BMI cohorts.
Quantitative US: Reproducibility of US Measurements (different sonographers) - Attenuation Coefficient (dB/cm-MHz) | Research visit 1 (up to 14 months)
  Biomarkers of liver steatosis are measured and analyzed for their reproducibility between different sonographers in the healthy BMI cohort.
Quantitative US: Reproducibility of US Measurements (different sonographers) - Backscatter Coefficient (1/cm*sr) | Research visit 1 (up to 14 months)
  Biomarkers of liver steatosis are measured and analyzed for their reproducibility between different sonographers in the healthy BMI cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Rosado-Mendez, PhD, Principal Investigator — University of Wisconsin, Madison; Diego Hernando, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No